CLINICAL TRIAL: NCT07296380
Title: Development of a Manual Therapy Application Behavior Scale Among Physiotherapists: A Validity and Reliability Study
Brief Title: Manual Therapy Behavior Scale in Physiotherapists
Status: Enrolling by invitation | Type: Observational
Sponsor: Uşak University (Other)
Collaborators: Pamukkale University (Other)
Responsible Party: Sponsor
Other Study IDs: E-60116787-020-789576
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Attitude of Health Personnel
Keywords: Physical Therapy Specialty; Attitude of Health Personnel; Clinical Competence; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Phsysiotherapists: Healthy adult physiotherapists who are actively working in public or private healthcare institutions or university clinics in Turkey and have received training or basic practical experience in manual therapy. Participation is voluntary, and no clinical intervention will be performed.

SUMMARY:
The aim of this study is to develop a scale to assess the manual therapy application behaviors of physiotherapists in Türkiye, based on the Theory of Planned Behavior (Ajzen, 1991). A literature-based item pool will be created, and expert opinion (Delphi method) will be obtained to ensure content validity. The final scale will be administered online to physiotherapists, and construct validity and reliability analyses will be conducted. The study aims to contribute scientifically to the determination of manual therapy application behaviors in physiotherapy practices, the understanding of clinical decision-making processes, and the measurement of behavioral intention. No risks were anticipated for the participants, and data collection was voluntary.

DETAILED DESCRIPTION:
Manual therapy is an evidence-based intervention method based on manual techniques widely used by physiotherapists in the treatment of musculoskeletal disorders. However, clinicians' decisions to implement manual therapy are influenced by multidimensional factors such as personal attitudes, professional beliefs, institutional policies, educational experiences, and the culture of clinical practice. The use of behavior-based theoretical models is recommended to evaluate these factors together.

The Theory of Planned Behavior (Ajzen, 1991) is a powerful approach that explains individuals' intentions to perform a specific behavior through variables such as attitude, subjective norm, perceived behavioral control, and intention. Although this theory is frequently used to understand the clinical decision-making processes of healthcare professionals, there is no valid and reliable measurement tool in Turkey for measuring behavior toward manual therapy practices.

This study will develop a new scale adapted to Turkish culture to assess physiotherapists' manual therapy practices in a theoretically based manner. The research will consist of three phases:

Item Development Phase:

The item pool generated through the literature review will be presented to expert physiotherapists.

Expert Panel/Delphi Phase:

Experts will evaluate the items based on content validity, and items will be revised or removed based on consensus. In this phase, the Content Validity Index (CVI) and Content Validity Ratio (CVR) will be evaluated.

Statistical Analysis Phase:

The final scale will be administered online to physical therapists.

ELIGIBILITY:
Inclusion Criteria:

* Be actively working as a physiotherapist in Turkey (public/private hospital, university hospital, private clinic, etc.)
* Have received basic training in manual therapy or have clinical practice experience
* Be a healthy adult aged 22 or over
* Be able to read and understand Turkish (the survey language is Turkish)
* Agree to participate in the study voluntarily and provide individual informed consent

Exclusion Criteria:

* Professionals working in healthcare fields other than physiotherapy
* Physiotherapists without manual therapy experience
* Participants who complete the survey form incompletely, incorrectly, inconsistently, or provide duplicate entries
* Individuals who refuse to provide informed consent
* Individuals who withdraw their voluntary consent during the research process

Ages: 22 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study population for this study consists of healthy adult physiotherapists actively working in public or private healthcare institutions or university hospitals in Turkey. Participants are expected to have basic training in manual therapy or clinical practice experience. Data collection will be conducted online, and participation is entirely voluntary. No medical interventions will be administered; data will be collected solely through a self-report questionnaire.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2026-03-25 (Estimated); Study Completion 2026-03-25 (Estimated)

PRIMARY OUTCOMES:
Manual Therapy Application Behavior Scale for Physiotherapists | One-time evaluation during the data collection period
  "Manual Therapy Application Behavior Scale in Physiotherapists" is a 7-point Likert-type (1 = Strongly disagree, 7 = Strongly agree) self-report scale developed based on Ajzen's Planned Behavior Theory. Higher scores reflect more positive attitudes, stronger subjective norms, higher perceived behavioral control, and higher behavioral intentions among physical therapists toward manual therapy. Construct validity will be assessed using internal consistency (Cronbach's alpha), item-total correlations, test-retest reliability, and confirmatory factor analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Because data is collected entirely on a voluntary basis, protecting participant privacy is a priority. Therefore, there are no plans to share Individual Participant Data (IPD) with third parties.